CLINICAL TRIAL: NCT04485988
Title: Influence of Beta Blockers on Prognosis in Patients With Acute Myocardial Infarction Complicated With Normal Ejection Fraction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dongying Zhang, Professor, Chongqing Medical University
Other Study IDs: 2020-06-25
Record Dates: First submitted 2020-07-22; First posted 2020-07-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: AMI
MeSH Terms: interventions — Adrenergic beta-Antagonists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No-beta blocker
- beta blocker
  Interventions: Drug: Beta blocker

INTERVENTIONS:
Drug: Beta blocker — Duration of medication
  Groups: beta blocker

SUMMARY:
To understand the effect of beta blockers on the prognosis of patients with acute myocardial infarction with preserved ejection fraction.

DETAILED DESCRIPTION:
The use of beta blockers is an important component of drug therapy for myocardial infarction, but in some exceptional cases, evidence-based evidence for their use is insufficient, and we seek to understand the prognostic impact of beta blockers on patients enrolled in long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute myocardial infarction

Exclusion Criteria:

* Previous history of heart failure admission Killip class > I class cancer pregnant

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The enrolled patients were from the First Affiliated Hospital of Chongqing Medical University, and the patient information was obtained from the medical record system
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2015-07-01 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Death | The median time of 3 years
  all-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: dongying zhang, doctor, Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China